CLINICAL TRIAL: NCT07373015
Title: Comparision of Safety and Efficacy Between Modified Double Snare Assisted EMR (mDS-EMR) and ESD for Rectal Neuroendocrine Tumors Smaller Than 1cm: a Prospective Non-inferiority Randomized Controlled Study
Brief Title: Modified Double Snare Assisted EMR (mDS-EMR) VS ESD for Rectal Neuroendocrine Tumors Smaller Than 1cm
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0755; 2025-LCYJ-MS-12 (Other Grant/Funding Number: the Affiliated Drum Tower Hospital of Nanjing University Medical School)
Record Dates: First submitted 2026-01-09; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Rectal Neuroendocrine Tumors
Keywords: Endoscopic Submucosal Dissection; Endoscopic Mucosal Resection; rectal neuroendocrine tumor
MeSH Terms: interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESD (Active Comparator): The traditional ESD treatment method is adopted, which includes submucosal injection of normal saline and methylene blue suspension, cutting and dissection by mucosal incision knife, hemostasis and cliping of the wound. Traction is allowed during the operation.
  Interventions: Procedure: endoscopic submucosal dissection
- mDS-EMR (Experimental): Modified double snare assisted EMR was used for treatment. Put the first snare for resecting outside the endoscope body. Then put the second snare at the base through the channel to tighten the lesion. Finally, place the first snare below the second one to tighten the lesion and perform electrically-assisted removal. Then, metal clips will be used to close the wound.
  Interventions: Procedure: modified double snare assisted endoscopic mucosal resection

INTERVENTIONS:
Procedure: modified double snare assisted endoscopic mucosal resection — A polypectomy snare (resection snare) was placed outside of the endoscope. After approaching the lesion, a second polypectomy snare (capture snare) was inserted through the biopsy channel of the endoscope to grasp and lift the lesion. The snare preloaded outside of the endoscope was released, passed through the capture snare and positioned below the capture snare to grasp the base of the lesion. Once the lesion was securely grasped, it was resected by resection snare to achieve en bloc resection. The wounds were closed by clips.
  Arms: mDS-EMR
Procedure: endoscopic submucosal dissection — The procedure includes submucosal injection of normal saline and methylene blue suspension, cutting and dissection by mucosal incision knife (such as Dual knife, Golden knife or Kunpeng knife, etc.) , hemostasis and sealing of the wound. Traction is allowed during the operation.
  Arms: ESD

SUMMARY:
The aim of this study is evaluating and safety and efficacy between the modified double snare EMR and ESD. It is intended to prove that for rectal neuroendocrine tumors within 1 cm, the complete resection rate of the mDS-EMR is not inferior to that of ESD, but may with shorter operation time, lower complication rate and lower treatment cost.

DETAILED DESCRIPTION:
A prospective, single-center, randomized controlled non-inferiority trial was designed to compare the safety and efficacy of modified double snare EMR (mDS-EMR) with endoscopic submucosal dissection (ESD) for the resection of rectal neuroendocrine tumors. The study have 4 main research contents. 1, Whether the resection effect of mDS-EMR is not inferior to that of ESD, and the treatment effect is evaluated by the complete resection rate (R0 resection rate). 2, Whether the operation time of mDS-EMR is significantly shorter than that of ESD. 3, To compare the safety between mDS-EMR and ESD, and whether the mDS-EMR can reduce the risk of intraoperative and postoperative adverse events. 4, To compare the postoperative hospital stay, surgical costs and hospitalization costs between mDS-EMR and ESD.

ELIGIBILITY:
Inclusion Criteria:

1. Typical rectal neuroendocrine tumors by endoscopy (within 15cm from the anal verge, yellowish subepithelial elevation with a smooth surface, and dilated blood vessels in some areas).
2. The maximum diameter of the lesion is smaller than 1cm by preoperative endoscopic assessment.
3. Lesion is located within the mucosal and submucosal layer by preoperative endoscopic assessment.
4. Patients can understand and sign the informed consent.

Exclusion Criteria:

1. Poor coagulation function(PT>15 seconds or APTT>45 seconds or INR>2.0)
2. With severe cardiovascular or cerebrovascular diseases and cannot tolerate operation( with a history of stroke or myocardial infarction within the past month or with severe heart failure and cardiac function grade III)
3. Indication of metastasis by preoperative imaging examinations
4. With more than or equal to 2 rectal neuroendocrine tumors
5. With other complications that are not suitable for this study by multidisciplinary team assesment
6. Cases of recurrence after operation for neuroendocrine tumors

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
complete resection | Day 30
  Rate of complete en bloc resection with microscopically negative margins.

SECONDARY OUTCOMES:
En bloc resection | Day 30
  Rate of complete resection as a single piece
operation success rate | Periprocedural
  Technical success was defined as the completion of procedure without abortion or conversion to other procedure
operation time | Periprocedural
  Operation time of ESD refers to the period from marking to completely removing the lesion, including submucosal injection, circumferential incision, submucosal dissection, additional submucosal injection and hemostasis during the operation and closure of the wound.
  Operation time of mDS-EMR refers to the period from the placing of the external snare to completely removing the lesion, hemostasis and closure of the wound.
Postoperative hospital stay | through study completion, an average of 30 days
  Period from the day of operation to discharge
operation-related expenses | through study completion, an average of 30 days
  Consumables cost of mDS-EMR and ESD
Average hospitalization expenses | through study completion, an average of 30 days
  All the expenses during the hospitalization period

OTHER OUTCOMES:
Delayed perforation | 30 days after the operation
  Postoperative abdominal pain, along with pelvic infection. Free gas in the pelvic cavity can be observed by imaging examination.
Delayed bleeding | 30 days after the operation
  Hemorrhage occurs withing 30 days after the procedure that requires endoscopic, radiological, or surgical intervention, or a blood transfusion may be required.
Intraoperative bleeding | Intraoperative
  arterial bleeding or active oozing for more than 30 seconds during the operation, which required endoscopic, radiological, or surgical intervention.
Intraoperative perforation | Intraoperative
  Damage of muscular layer of rectal wall and a hole to extracavitary tissue can be observed by endoscopy.